CLINICAL TRIAL: NCT05080647
Title: Examining the Impacts of Parent Mightier Play as a Supplement to Child Mightier Play
Brief Title: Examining the Impacts of Parent Mightier Play
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neuromotion Labs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 995MIGH21
Record Dates: First submitted 2021-09-28; First posted 2021-10-18 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2021-10

CONDITIONS: Emotional Regulation
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mightier Child Play (Active Comparator): 8 weeks of use ad-libitum. Parents will be encouraged to have their children play Mightier games at least 3 times a week (totalling 45 minutes or more play each week) for the 8-week duration. Parents in the Child Play condition will be advised specifically to not play Mightier for the 8-week duration of the study.
  Interventions: Behavioral: Mightier online gameplay
- Mightier Child and Parent Play (Experimental): 8 weeks of use ad-libitum. Parents will be encouraged to have their children play Mightier games at least 3 times a week (totalling 45 minutes or more of play each week) for the 8-week duration. Additionally, parents in the Child and Parent Play condition will be encouraged to play Mightier games at least once a week (totalling 15 minutes or more of play each week) for the 8-week duration.
  Interventions: Behavioral: Mightier online gameplay

INTERVENTIONS:
Behavioral: Mightier online gameplay — Mightier is a video-game-based biofeedback intervention that capitalizes on children's love of video games to increase emotional awareness and facilitate emotion regulation practice through heart rate (HR) control. Each family receives a Mightier Kit (Mighty Band heart rate monitor, dedicated Mightier tablet unless the family prefers to use their own device) and the Mightier App. Children wear a "Mighty Band" heart rate monitor on their arm while they play any one of 26+ games. As their heart rate rises the games become more difficult. For example, during a cooking game, smoke may appear on the screen and obscure the player's view. Children can either opt into an explicit cool down activity (deep breathing, progressive muscle relaxation, crossing the midline, or visualization) or cool down on their own. By simply playing Mightier, children are motivated to practice calming strategies in moments of challenge.
  Other Names: Mightier

SUMMARY:
A randomized controlled trial comparing a group in which only child participants play Mightier video games for 8 weeks (Child Play group) to a group in which child and parent participants play Mightier video games for 8 weeks (Child and Parent Play group).

DETAILED DESCRIPTION:
Mightier is a mobile app-based biofeedback video game platform that facilitates emotion regulation skill-building among children ages 6-14. The technology behind Mightier's mobile app has been validated in two independent sham-controlled randomized controlled trials, where the investigators have seen decreases in clinical symptoms of aggression and disruptive behaviors, as well as lowered family stress without adverse events.

The study utilizes a parallel randomized controlled design comparing groups of participant families whose children play Mightier video games without parent play to groups of participant families in which both children and parents play Mightier video games. Self-report measures will be completed by participant children and parents.

The study consists of three primary phases: Pre-Study, Active Engagement, and Follow-Up. During the Pre-Study Phase, participants will undergo pre-screening and screening to evaluate interest and eligibility for the study, and participants who consent to participate in the study will complete baseline measures and be randomized into treatment groups. Mightier games will be shipped to participants during or shortly after their Pre-Study call. Participants will be instructed to begin Mightier gameplay as soon as Mightier games arrive at their homes, which will begin the Active Engagement Phase of the study.

During the 8-week Active Engagement Phase, participants will be encouraged to play Mightier games in a way that corresponds to their study condition, and they will be offered engagement support in the form of brief weekly check-ins.

After completion of the Active phase, participants will have a brief Follow-up phase, consisting of one video call during which child and parent participants will complete self-report follow-up measures.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-12 at the time of screening
* Regular access to WiFi (for Mightier gameplay device connection)

Exclusion Criteria:

* Prior Mightier use
* Diagnosed Intellectual Disability (by history)
* Planned medication changes during the 8-week study period

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-03-19 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Change in child behavior and emotion problems measured on BFS at Week 8 | Baseline and Week 8
  Behavior and Feelings Survey (BFS): The BFS (Weisz et al., 2014) is a 12-item scale measuring child behavior and emotion problems. The child's parent is prompted to read the survey questions to the child and to note the child's responses. The researcher will screen share the BFS form and record child responses in the form. Children will complete the BSF at baseline and Week 8. Items are rated on a scale from 0 (not a problem) to 4 (a very big problem). Three scale scores can be derived: Internalizing Problems (sum of items 1-6), Externalizing Problems (sum of items 7-12), and Total Problems (sum of items 1-12).
Change in child irritability from baseline measured on ARI-P at Week 8 | Baseline and Week 8
  Affective Reactivity Index-Parent Report (ARI-P): The ARI is a 7-item scale that consists of 6 symptom items and 1 impairment item. The scale was designed to determine irritable mood rather than behavioral consequences such as hostility and acts of aggression (Stringaris et al., 2012). The individual items are scored 0,1, 2, and only the first six items are summed to form the total score, with a minimum score of 0 and a maximum score of 18, and higher scores indicating greater severity of irritability symptoms. The seventh item is an impairment item and it is analysed separately, with a minimum score of 0 and a maximum score of 3, and higher scores indicating greater irritability symptom severity. Parent participants will complete the ARI-P at baseline and Week 8.
Parent perception of change in child emotion regulation from baseline measured on GIS at Week 8 | Baseline and Week 8
  Global Improvement Scale (GIS): The GIS is a parent self-report question that asks parents if they have noticed any overall improvements in their child's emotion regulation, with response options ranging from (1) very much improved to (7) very much worse. Minimum score = 1, Maximum score = 7, with higher numbers indicating less improvement, or worsening. The GIS has not been scientifically validated. Parent participants will complete the GIS at Week 8.

SECONDARY OUTCOMES:
Change in parent emotion regulation from baseline measured on DERS-18 at Week 8 | Baseline and Week 8
  Difficulties in Emotion Regulation Scale, 18-question short form (DERS-18): The DERS-18 (Victor & Klonsky, 2016) is an 18-question measure of the respondent's emotion regulation experiences. For scoring, three responses are reverse-coded then all responses are summed, resulting in an overall score and scores on 6 subscales: Awareness, Clarity, Goals, Impulse, Nonacceptance, and Strategies. Higher scores indicate greater emotion regulation difficulties. Parent participants will complete the DERS-18 at baseline and Week 8.
Change in parent beliefs about intervention credibility and effectiveness from baseline, measured on the CEQ-P at Week 4 and Week 8 | Baseline, Week 4, and Week 8
  Credibility and Expectancies Questionnaire - Parent Version (CEQ-P): Parent participants will respond to the CEQ-P (Nock et al., 2007), a 6-question assessment of their beliefs about credibility and effectiveness of the intervention, at baseline, Week 4, and Week 8. Items 1, 2, 3, and 5 are scored on a nine-point scale (1 = not a lot / not much; 9 = a lot / very much). Items 4 and 6 are scored on an 11-point scale (e.g., 0-100%), then recoded for scoring to correspond to the 1-9 point scale used for items 1-3 and 5, collapsing the values from 40-60% into one value, 5.
Change in child-parent relationship from baseline, measured on the CPRS-SF at Week 8 | Baseline and Week 8
  Child-Parent Relationship Scale (CPRS-SF): The CPRS-SF (Pianta, 1992) is a 15-item self-report instrument completed by parents that assesses their perceptions of their relationship with their child. The 15 items are rated on 5-point Likert scales. It is applicable to children ages 3-12. The CPRS-SF is scored in two subscales: an 8-item Conflict subscale (minimum score = 8, maximum score = 40, higher score indicates greater conflict), and a 7-item Closeness subscale (minimum score = 7, maximum score = 35, with greater score indicating greater closeness). Parent participants will complete the CPRS-SF at baseline and Week 8.

CONTACTS AND LOCATIONS:
Locations (1):
- Neuromotion Labs, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Only Mightier research staff will have access to individual participant data, including family demographics data and data from child and parent self-report measures.

REFERENCES:
- [Background] RC Pianta - Unpublished measure, University of Virginia, 1992
- [Background] Stringaris A, Goodman R, Ferdinando S, Razdan V, Muhrer E, Leibenluft E, Brotman MA. The Affective Reactivity Index: a concise irritability scale for clinical and research settings. J Child Psychol Psychiatry. 2012 Nov;53(11):1109-17. doi: 10.1111/j.1469-7610.2012.02561.x. Epub 2012 May 10. PMID 22574736
- [Background] Weisz JR, Vaughn-Coaxum RA, Evans SC, Thomassin K, Hersh J, Ng MY, Lau N, Lee EH, Raftery-Helmer JN, Mair P. Efficient Monitoring of Treatment Response during Youth Psychotherapy: The Behavior and Feelings Survey. J Clin Child Adolesc Psychol. 2020 Nov-Dec;49(6):737-751. doi: 10.1080/15374416.2018.1547973. Epub 2019 Jan 18. PMID 30657721
- [Background] Nock, M.K., Ferriter, C. & Holmberg, E. Parent Beliefs about Treatment Credibility and Effectiveness: Assessment and Relation to Subsequent Treatment Participation. J Child Fam Stud 16, 27-38 (2007). https://doi.org/10.1007/s10826-006-9064-7
- [Background] Victor, S.E., Klonsky, E.D. Validation of a Brief Version of the Difficulties in Emotion Regulation Scale (DERS-18) in Five Samples. J Psychopathol Behav Assess 38, 582-589 (2016). https://doi.org/10.1007/s10862-016-9547-9